CLINICAL TRIAL: NCT02407938
Title: Normal Values for Esophageal High Resolution Manometry in an Advanced Protocol Using a Test Meal
Brief Title: Normal Values for Esophageal High Resolution Manometry in an Advanced Protocol Including Liquid Swallows and a Solid Test Meal
Acronym: Rice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KEK-ZH-Nr. 2013-0176
Record Dates: First submitted 2015-03-18; First posted 2015-04-03 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: dysphagia; reflux symptoms; retrosternal pain
MeSH Terms: conditions — Deglutition Disorders | interventions — Flour

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rice meal (Experimental): High resolution manometry will be performed. Esophageal function will be tested using liquid swallows, solid swallows and a test meal (200g rice)
  Interventions: Other: Rice meal

INTERVENTIONS:
Other: Rice meal

SUMMARY:
Normal values for measurements of high resolution manometry in a protocol which includes isolated liquid swallows in upright and recumbent position, free drinking of water, a solid test meal and a postprandial observational period will be determined.

DETAILED DESCRIPTION:
The investigators will recruit healthy volunteers and ask for study participation. After providing informed consent, participants will be questioned using standardized questionnaires assessing symptoms of reflux, dysphagia, gastrointestinal symptom burden and depression. Participants will be tested using our advanced protocol for high resolution esophageal manometry. This protocol includes individual liquid swallows, free drinking of water, a standardized test meal (200g rice) and a postprandial observational period. Normal values for liquid and solid swallows will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers without gastrointestinal co-morbidity

Exclusion Criteria:

* Inability or unwillingness to provide informed consent
* Any relevant current or past gastrointestinal morbidity (including diseases relevant previous surgery).
* Relevant gastrointestinal symptoms
* Relevant medication (as specified below) within the last 4 weeks
* Age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Values for HRM data (IRP, DCI, DL) in healthy volunteers | 1 hour
  Normal values for measurements of high resolution manometry in a protocol which includes isolated liquid swallows in upright and recumbent position, free drinking of water, a solid test meal

SECONDARY OUTCOMES:
discomfort on a VAS from 1-10 for each type of measurement | 1 hour
  Discomfort during different steps of the investigation

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Ang D, Misselwitz B, Hollenstein M, Knowles K, Wright J, Tucker E, Sweis R, Fox M. Diagnostic yield of high-resolution manometry with a solid test meal for clinically relevant, symptomatic oesophageal motility disorders: serial diagnostic study. Lancet Gastroenterol Hepatol. 2017 Sep;2(9):654-661. doi: 10.1016/S2468-1253(17)30148-6. Epub 2017 Jul 3. PMID 28684262
- [Derived] Hollenstein M, Thwaites P, Butikofer S, Heinrich H, Sauter M, Ulmer I, Pohl D, Ang D, Eberli D, Schwizer W, Fried M, Distler O, Fox M, Misselwitz B. Pharyngeal swallowing and oesophageal motility during a solid meal test: a prospective study in healthy volunteers and patients with major motility disorders. Lancet Gastroenterol Hepatol. 2017 Sep;2(9):644-653. doi: 10.1016/S2468-1253(17)30151-6. Epub 2017 Jul 3. PMID 28684261